CLINICAL TRIAL: NCT06092047
Title: Clinical Study of Universal Off-the-shelf Cell Products in Patients With CD19-positive Relapsed/Refractory B-cell Hematolymphatic Malignancies.
Brief Title: UTAA09 Injection in the Treatment of Relapsed/Refractory Hematolymphatic Malignancies.
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Collaborators: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-CART-UTAA09-001
Record Dates: First submitted 2023-10-07; First posted 2023-10-23 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-05

CONDITIONS: CD19-positive Relapsed or Refractory B-cell Malignancies
Keywords: CD19 target; UCAR-T
MeSH Terms: interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: UTAA09 injection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- UTAA09 cells for infusion (Experimental): Off-the-shelf γδT cells with a CD19-redirected Chimeric Antigen Receptor. Route of administration: Intravenous injection. Lymphodepleting conditioning regimen: A combination of fludarabine and cyclophosphamide will be administered at Day-7~Day-2.
  Interventions: Biological: UTAA09 cells for infusion; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: UTAA09 cells for infusion — Intravenous injection, dosage:1-10×10^8 CAR+ γδT cells, Cell concentration: 2×10^7 cells/mL.
Drug: Fludarabine — 30 mg/m^2/day×4 days
Drug: Cyclophosphamide — 1000 mg/m^2/day×3 days

SUMMARY:
This study is designed for exploring the preliminary safety and efficacy of the recombinant allogeneic healthy γδT cells transduced with the anti-CD19 lentiviral vector in patients with CD19-positive B cell hematolymphatic malignancies.

DETAILED DESCRIPTION:
A single arm open-label clinical study is designed to prelinarily determine the safety, efficacy, the ratio of CD19-positive cells in peripheral blood and cell kinetics after administration of UTAA09 injection in patients with CD19-positive relapsed/refractory B-cell hematolymphatic malignancies. All subjects will receive UTAA09 cells infusion.

Primary objective: explore the preliminary safety and efficacy of UTAA09 injection in patients with CD19-positive relapsed/refractory B-cell line hematolymphatic malignancies.

Secondary objectives:

1. explore the distribution, amplification and survival of UTAA09 cells in vivo after administration of UTAA09 injection;
2. explore the ratio of CD19-positive cells in peripheral blood after administration of UTAA09 injection.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 3~70 (including cut-off values), regardless of gender and race;
2. Expected survival time>12 weeks;
3. ECOG score 0-2;
4. CD19-positive relapsed/refractory B-cell hematolymphatic malignancies;
5. Liver and kidney function, cardiopulmonary function meet the following requirements:

   1. Creatinine ≤ 1.5 ULN;
   2. Left ventricular ejection fraction ≥ 45%;
   3. blood oxygen saturation>91%;
   4. Total bilirubin ≤ 1.5 × ULN； ALT and AST ≤ 2.5 × ULN;
6. Be able to understand the trial and have signed the informed consent.

Exclusion Criteria:

1. Those with graft-versus-host disease (GVHD) or requiring long-term systemic immunosuppressants;
2. Malignant tumors other than CD19-positive hematologic malignancies within 5 years prior to screening, except adequately treated cervical carcinoma in situ, basal cell or squamous epithelial cell skin cancer, local prostate cancer after radical resection, and breast ductal carcinoma in situ after radical resection;
3. Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and peripheral blood hepatitis B virus (HBV) DNA titer outside the normal reference range; Those who are positive for hepatitis C virus (HCV) antibodies and positive for hepatitis C virus (HCV) RNA in peripheral blood; Human immunodeficiency virus (HIV) antibody positive person; Positive for cytomegalovirus (CMV) DNA testing; those who test positive for syphilis;
4. Serious heart disease: including but not limited to unstable angina, myocardial infarction (within 6 months before screening), congestive heart failure (NYHA classification ≥ III), and serious arrhythmia;
5. Unstable systemic diseases judged by the investigator: including but not limited to severe liver, kidney or metabolic diseases requiring drug treatment;
6. Within 7 days before screening, there is active infection or uncontrollable infection requiring systemic treatment (except for mild genitourinary system infection and upper respiratory tract infection);
7. Pregnant or lactating women, female subjects who planned to conceive within 1 year of cell infusion or male subjects whose partner planned pregnancy within 1 year of their cell infusion;
8. Screening participants (except for inhalation or local use) who were receiving systemic steroid treatment within 7 days before screening or who were judged by the investigator to require long-term systemic steroid therapy during treatment;
9. Participated in other clinical studies within 3 month before screening;
10. There was evidence of central nervous system involvement at participant screening;
11. Conditions that the investigators considered unsuitable for enrollment.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Assessment of the safety after UTAA09 injection treatment | About 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.
Evaluation of the efficacy after UTAA09 injection treatment | About 3 months
  3-month total response rate (ORR) which includes CR, CRi, and PR will be assessed.

SECONDARY OUTCOMES:
Assessment of pharmacokinetic (about Cmax) | About 2 years
  Assessment of the peak Plasma Concentration (Cmax) of UTAA09 cells amplified in peripheral blood after administration.
Assessment of pharmacokinetic (about Tmax) | About 2 years
  Assessment of the time to reach the highest concentration (Tmax) of UTAA09 cells amplified in peripheral blood after administration.
Assessment of pharmacokinetic (about AUC0-28d) | About 2 years
  Assessment of the Area under the plasma concentration versus time curve (AUC) for 28 days after UTAA09 cells administration.
Assessment of pharmacokinetic (about AUC0-90d) | About 2 years
  Assessment of the Area under the plasma concentration versus time curve (AUC) for 90 days after UTAA09 cells administration.
Evaluation of Pharmacodynamic | About 2 years
  To determine the depletion of peripheral blood CD19-positive B cells at each time point, the concentration of CAR-γδT-associated serum cytokine (CRP, IL-6, etc.).
To evaluate the efficacy (Overall Survival) | About 2 years
  Defined as the time from the start of UTAA09 injection therapy to patient death (due to any cause).
To evaluate the efficacy (Duration Of Response) | About 2 years
  Defined as the time from the first tumor assessment of CR or PR, CR or CRi to the first assessment of disease recurrence or progression or death (due to any cause).
To evaluate the efficacy (Progression Free Survival) | About 2 years
  Defined as the time from the start of UTAA09 injection therapy to the first disease progression or recurrence or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xingbing Wang, MD, Principal Investigator — The First Affiliated Hospital of USTC (Anhui Provincial Hospital)
Locations (1):
- The First Affiliated Hospital of USTC (AnHui Provincial Hospital), Hefei, Anhui, China